CLINICAL TRIAL: NCT00250848
Title: Lung Cancer Case Registry and Tissue Resource
Status: Terminated | Type: Observational
Why Stopped: This is not a clinical trial and was inadvertently entered into the system.
Sponsor: University of New Mexico (Other)
Responsible Party: Sponsor
Other Study IDs: 2903C
Record Dates: First submitted 2005-11-04; First posted 2005-11-08 (Estimated); Last update posted 2024-01-08 (Actual); Status verified 2024-01

CONDITIONS: Lung Cancer
Keywords: Lung Diseases; Cancer
MeSH Terms: conditions — Lung Neoplasms; Lung Diseases; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Blood samples, and sputum (phlegm) samples.
Oversight: Data Monitoring Committee: No

SUMMARY:
Potential participants in the Lung Cancer Case Registry will be all patients diagnosed or evaluated for possible treatment of lung cancer at the Cancer Research and Treatment Center (CRTC) and New Mexico Veterans Health Care System (NMVHCS).

DETAILED DESCRIPTION:
Lung cancer is the most common cause of cancer death in the US in both men and women. This research study will enroll lung cancer patients into a registry to study changes in DNA (or genetic material) that may be associated with development of lung cancer or other lung diseases such as chronic obstructive pulmonary disease (COPD). We will also study the role of eating habits on lung cancer diagnosis and treatment, as well as the effects of the disease and treatment on quality of patient's lives.

ELIGIBILITY:
Inclusion Criteria:

* Potential participants in the Lung Cancer Case Registry will be all patients diagnosed or evaluated for possible treatment of lung cancer at the CRTC and NMVHCS. Recruiting will primarily be performed through the Multidisciplinary Chest Clinics held weekly at each hospital. These clinics are staffed by the Principal Investigator (PI) and Reza Mehran, MD, a thoracic surgeon at both hospitals and a co-investigator on this submission. Approximately 90% of all lung cancer cases diagnosed at the NMVHCS, and a somewhat smaller proportion of cases treated in the Cancer Center, are seen in these clinics. Additional cases will be identified through review of new patient visits to each hospital with a diagnosis of lung cancer; Drs. Crowell and Mehran also maintain weekly contact with pathology and oncology services at both facilities, which will facilitate case identification at NMVHCS and University Hospital. Finally, patient contact records will be correlated with tumor registry records at both hospitals, which will identify any cases not captured through the above mechanisms. Although these cases may be identified several weeks after initial diagnosis, all attempts will still be made to contact the patient and family for enrollment into the registry. Most Spanish-speaking patients served by the CRTC and the NMVHCS are bilingual, and a language barrier has not been a problem in other similar studies conducted by the PI. However, Spanish-speaking personnel are available to obtain consent and answer any questions if necessary.

Exclusion Criteria:

* Patients will be excluded if they cannot provide written informed consent.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients (male or female) with Lung cancer.
Sampling Method: Probability Sample
Enrollment: 750 (Actual)
Dates: Start 2004-03 (Actual); Primary Completion 2015-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
DNA Change | one year

CONTACTS AND LOCATIONS:
Overall Officials: Richard Crowell, MD, Principal Investigator — University of New Mexico
Locations (2):
- United States (2):
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - New Mexico Veterans Administration Health Care System, Albuquerque, New Mexico